CLINICAL TRIAL: NCT04608617
Title: Observational Study of Automated Detection for Identification, Triage, and Timely Intervention in Large Vessel Occlusions- SYNCHRONISE
Brief Title: SYNCHRONISE: LVO Triage Timing and Outcome Study
Status: Completed | Type: Observational
Sponsor: Viz.ai, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VIZ-LVO-03
Record Dates: First submitted 2020-10-11; First posted 2020-10-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke, Ischemic
Keywords: Artificial Intelligence; Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pre-Viz: Pre-Viz LVO implementation patient data utilized as a control data set
  Interventions: Other: Baseline Effectiveness Cohort
- Post-Viz: Patient data collected post-Viz LVO implementation
  Interventions: Device: Viz LVO (De Novo Number DEN170073)

INTERVENTIONS:
Device: Viz LVO (De Novo Number DEN170073) — Viz LVO is a notification-only, parallel workflow tool for use by hospital networks and trained clinicians to identify and communicate images of specific patients to a specialist, independent of standard of care workflow.
  Viz LVO uses an artificial intelligence algorithm to analyze images for findings suggestive of a pre-specified clinical condition and to notify an appropriate medical specialist of these findings in parallel to standard of care image interpretation. Identification of suspected findings is not for diagnostic use beyond notification. Specifically, the device analyzes CT angiogram images of the brain acquired in the acute setting and sends notifications to a neurovascular specialist that a suspected large vessel occlusion has been identified and recommends review of those images. Images can be previewed through a mobile application.
  Other Names: ContaCT
  Groups: Post-Viz
Other: Baseline Effectiveness Cohort — No Intervention was performed for the pre-Viz group. Record review to establish operational metrics only occurred.
  Groups: Pre-Viz

SUMMARY:
The objective of this study is to evaluate the impact of Viz LVO in hospital systems with non-interventional and interventional (spoke and hub) stroke centers on the timing and outcomes of patients with suspected acute ischemic stroke indicated for mechanical thrombectomy.

DETAILED DESCRIPTION:
This is a multi-center, non-randomized observational study of acute ischemic stroke patients whose CTA scans are analyzed by Viz LVO to support clinicians in making stroke triage decisions,. The study results will be compared to a cohort from enrolling centers prior to Viz LVO implementation that will serve as a historical control. Data will be collected retrospectively from the time of presentation through 90 days post discharge.

The study will include patients undergoing imaging for a suspected LVO acute ischemic stroke. The post-Viz LVO intervention group will consist of patients who either presented to or underwent transfer to an interventional center, from a non-interventional center, following image analysis by Viz LVO. Data will be collected retrospectively on consecutive patients meeting eligibility criteria from the date of implementation up to 5 years post implementation.

The control group will consist of patients who either presented to or underwent transfer to an interventional center, from a non-interventional center, for evaluation prior to the implementation of Viz LVO. Data will be collected on consecutive patients from one day prior to implementation, back as far as 2 years prior to implementation

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or greater
* Signs and symptoms consistent with the diagnosis of a large vessel occlusive stroke
* Pre-treatment National Institutes of Health Stroke Scale (NIHSS) ≥ 6
* Aspects Score ≥6
* Patient must have a suspected LVO in M1.
* Patient with an intention to treat with mechanical thrombectomy with confirmation of LVO by the CT/CTA radiographic report with the reading diagnosis.

Exclusion Criteria:

* Unable to undergo a brain imaging (i.e. severe contrast medium allergy, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients, that meet eligibility criteria, undergoing imaging for a suspected LVO acute ischemic stroke indicated for mechanical thrombectomy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Transfer patients: Time from spoke CT/CTA to door-out | up to 1 day (1440 minutes)
  Time in minutes from CT/CTA imaging to time leaving the spoke center
Non-transfer patients: Time from Hub door to groin puncture | up to 1 day (1440 minutes)
  Time in minutes from arrival a hub center to start time of treatment

SECONDARY OUTCOMES:
Time from Spoke Door-In to Door-Out (DIDO) | up to 1 day (1440 minutes)
  Time in minutes from arrival at spoke hospital to departure to hub hospital
Time from Spoke CT/CTA to Specialist Notification | up to 1 day (1440 minutes)
  Time in minutes from CT/CTA imaging to time an interventionalist was notified
Time from Spoke CT/CTA to Groin Puncture | up to 1 day (1440 minutes)
  Time in minutes from CT/CTA imaging to start time of treatment
Time from Spoke Door to Groin Puncture | up to 1 day (1440 minutes)
  Time in minutes from departure to hub hospital to start time of treatment
Length of ICU Stay/Total Length of Stay | Hospital admit to discharge, up to 30 days
  Number of days in hospital in the ICU and the total number of days in hospital
Modified Rankin Scale (mRS) at Discharge and 90 Days | 90 days
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. A score of 0 is a patient with no residual symptoms. Scores increase with severity to 5 which equals severe disability.
National Institutes of Health Stroke Scale (NIHSS) at Discharge | On date of discharge, up to 30 days
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored on a 3- to 5-point scale, with 0 as normal, and there is an allowance for untestable items. Scores range from 0 to 42, with higher scores indicating greater severity.
Patient Disposition at Discharge and 90 Days | 90 days
  Data will be collected on whether or not the patient was discharged to their home or another type of care facility, and where they are located 90 days post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Thomas Devlin, Principal Investigator — CHI Memorial; Dr. Ameer Hassan, Principal Investigator — Valley Baptist
Locations (3):
- United States (3):
  - Wellstar Neurosurgery, Atlanta, Georgia
  - Semmes-Murphey, Memphis, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas

IPD SHARING:
Plan to Share IPD: No